CLINICAL TRIAL: NCT07220785
Title: A Two-Part, Randomized, Placebo-Controlled Phase 3 Study of the Efficacy, Safety, and Pharmacokinetics of Mibavademab in Patients With Generalized Lipodystrophy
Brief Title: Efficacy and Safety of Mibavademab in Adult and Pediatric Patients With Generalized Lipodystrophy
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R4461-GLD-2285; 2024-519879-25-00 (Registry Identifier: EUCT Number)
Record Dates: First submitted 2025-10-22; First posted 2025-10-24 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Generalized Lipodystrophy
Keywords: Subcutaneous (SC) adipose tissue; GLD; Berardinelli-Seip Syndrome; Congenital Generalized Lipodystrophy; CGL; Lawrence Syndrome; Acquired Generalized Lipodystrophy; AGL
MeSH Terms: conditions — Lipodystrophy, Congenital Generalized; Lipodystrophy, Familial Partial

STUDY DESIGN:
Intervention Model Description: Part A will be double blinded; Part B will be open label
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part A: Arm A (Experimental)
  Interventions: Drug: Mibavademab
- Part A: Arm B (Experimental)
  Interventions: Drug: Mibavademab; Drug: Placebo
- Part A: Arm C (Experimental)
  Interventions: Drug: Mibavademab
- Part A: Arm D (Placebo Comparator)
  Interventions: Drug: Placebo
- Part B (Experimental)
  Interventions: Drug: Mibavademab

INTERVENTIONS:
Drug: Mibavademab — Administered as per the protocol
  Other Names: REGN4461
  Arms: Part A: Arm A; Part A: Arm B; Part A: Arm C; Part B
Drug: Placebo — Administered as per the protocol
  Arms: Part A: Arm B; Part A: Arm D

SUMMARY:
This study is researching a new drug called mibavademab (called "study drug"). The study involves participants with a condition called Generalized Lipodystrophy (GLD). The aim of the study is to see how well mibavademab works and what side effects it has. Researchers will also look at how much mibavademab is in the body at different times.

This is a 2-part study: Part A is an efficacy study in pediatric and adult participants, Part B is a safety and pharmacokinetic study in pediatric participants.

The study is researching several other questions, including:

* How mibavademab affects the amount of sugar in the blood
* How mibavademab affects the amount of fat (triglycerides) in the blood
* How mibavademab affects the amount of fat that has built up in the liver
* Whether the body makes antibodies against the study drug (which could make the drug less effective or could lead to side effects)

ELIGIBILITY:
Key Inclusion Criteria:

1. Diagnosis of congenital or acquired GLD as defined by Multi-Society Practice Guidelines

For Part A only:

1. Participants ≥2 years of age at screening
2. At least one of the below criteria are fulfilled during screening (measurements can be repeated once during screening period)

   * HbA1c ≥7%
   * Fasting TG ≥500 mg/dL
   * Fasting TG value of ≥300 mg/dL and the presence of another complication of GLD consistent with leptin deficiency (history of diabetes mellitus, hyperphagia, Metabolic Associated Fatty Liver Disease (MAFLD), polycystic ovary syndrome, etc)
3. Weight ≥15 kg at screening
4. Willing and able to provide, or have the treating physician provide, values of HbA1c and fasting TG from at least 6 months prior to screening, as described in the protocol

For Part B only:

1. Participants ≥2 and <12 years of age at screening
2. No metabolic criteria or minimum weight for study entry is required

Key Exclusion Criteria:

1. Has a current diagnosis of familial or acquired partial lipodystrophy or autoimmune (Type 1) diabetes mellitus
2. Any malignancy, eg, lymphoma, within the past 1 year, prior to screening visit, as described in the protocol
3. eGFR of <30 mL/min/1.73 m2 based on Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) creatinine or Schwartz equation, as applicable, at screening. Assessment can be repeated once
4. History of heart failure hospitalization, diagnosis of a myocardial infarction, stroke, clinically significant arrhythmia, as described in the protocol
5. Treatment with over-the-counter or prescription medications with the intention of weight loss within 3 months prior to the screening visit

For Part A only:

1. Treatment with metreleptin within 3 months of the screening visit
2. Addition or discontinuation of prescription medications or over-the-counter supplements for diabetes and/or dyslipidemia within 3 months prior to the start of the screening period, or changes in the use of these medications, as described in the protocol
3. Significant changes to lifestyle and diet, as described in the protocol
4. Current chronic treatment with high-dose corticosteroids, defined as use of higher than physiologic doses, as described in the protocol

NOTE: Other protocol defined inclusion/exclusion criteria apply.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2026-02-27 (Estimated); Primary Completion 2028-05-19 (Estimated); Study Completion 2028-09-08 (Estimated)

PRIMARY OUTCOMES:
Change in Hemoglobin A1c (HbA1c) | Through 36 weeks of exposure to mibavademab
  Part A
Percent change in fasting Triglycerides (TG) | Through 36 weeks of exposure to mibavademab
  Part A
Occurrence of Treatment Emergent Adverse Events (TEAEs) | Up to 15 months
  Part B
Severity of TEAEs | Up to 15 months
  Part B
Concentrations of total mibavademab in serum | Up to 15 months
  Part B

SECONDARY OUTCOMES:
Change in HbA1c compared to placebo | From baseline to week 20
  Part A
Change in HbA1c compared to placebo | From week 56 to week 64
  Part A
Change in HbA1c | From baseline to week 52
  Part B
Percent change in fasting TG compared to placebo | From baseline to week 20
  Part A
Percent change in fasting TG compared to placebo | From week 56 to week 64
  Part A
Percent change in fasting TG | From baseline to week 52
  Part B
Occurrence of HbA1c <7% | At week 20
  Part A
Occurrence of HbA1c <7% | Through 36 weeks of exposure to mibavademab
  Part A
Occurrence of HbA1c <6.5% | At week 20
  Part A
Occurrence of HbA1c <6.5% | Through 36 weeks of exposure to mibavademab
  Part A
Occurrence of fasting TG <500 mg/dL | At week 20
  Part A
Occurrence of fasting TG <500 mg/dL | Through 36 weeks of exposure to mibavademab
  Part A
Occurrence of fasting TG <200 mg/dL | At week 20
  Part A
Occurrence of fasting TG <200 mg/dL | Through 36 weeks of exposure to mibavademab
  Part A
Occurrence of fasting TG <150 mg/dL | At week 20
  Part A
Occurrence of fasting TG <150 mg/dL | Through 36 weeks of exposure to mibavademab
  Part A
Percent change in Liver Fat Content (LFC) | From baseline to week 20
  Part A
Percent change in Liver Fat Content (LFC) | From pre-mibavademab exposure to week 56
  Part A
Change in liver volume | From baseline to week 20
  Part A
Change in liver volume | From pre-mibavademab exposure to week 56
  Part A
Change in fasting glucose | From baseline to week 20
  Part A
Change in fasting glucose | Through 36 weeks of exposure to mibavademab
  Part A
Change in fasting glucose | From week 56 to week 64
  Part A
Change in total daily insulin dose | From baseline to week 20
  Part A
Change in total daily insulin dose | Through 36 weeks of exposure to mibavademab
  Part A
Change in total daily insulin dose | From week 56 to week 64
  Part A
Change in total daily insulin dose | From baseline to week 52
  Part B
Concentrations of total mibavademab in serum | Through Week 72
  Part A
Occurrence of anti-drug antibodies (ADA) to mibavademab | Through Week 72
  Part A
Occurrence of ADA to mibavademab | Through Week 60
  Part B
Titer of ADA to mibavademab | Through Week 72
  Part A
Titer of ADA to mibavademab | Through Week 60
  Part B
Occurrence of TEAEs | Through Week 72
  Part A
Severity of TEAEs | Through Week 72
  Part A

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/